CLINICAL TRIAL: NCT01738243
Title: Phase IV Study of Hyaluronic Acid Gels for Upper Lid Retraction in Active Stage Thyroid Eye Disease
Brief Title: Hyaluronic Acid Gels for Upper Lid Retraction in Active Stage Thyroid Eye Disease
Acronym: HALR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment challenges
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Rootman, Clinical Instructor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRE#12-003174
Record Dates: First submitted 2012-10-06; First posted 2012-11-30 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Thyroid Eye Disease
Keywords: Thyroid; Thyroid Eye Disease; Thyroid Orbitopathy; Eyelid Retraction; Upper Eyelid Retraction
MeSH Terms: conditions — Graves Ophthalmopathy; Thyroid Diseases | interventions — Restylane; belotero balance; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unilateral Upper Eyelid Retraction (Experimental): This arm will consist of participants with unilateral upper eye lid retraction secondary to thyroid eye disease (TED).
  Patients enrolled will be randomized 1:1 to Hyaluronic Acid Gel Injection or Saline injection
  Interventions: Drug: Hyaluronic Acid Gel injection; Drug: Saline injection
- Bilateral Upper Eyelid Retraction (Experimental): This arm will consist of participants with bilateral upper eye lid retraction secondary to thyroid eye disease (TED).
  Patients enrolled will be randomized 1:1 to Hyaluronic Acid Gel injection or Saline injection
  Interventions: Drug: Hyaluronic Acid Gel injection; Drug: Saline injection

INTERVENTIONS:
Drug: Hyaluronic Acid Gel injection — The conjunctiva is anesthetized with Proparacaine Hydrochloride Ophthalmic Solution, 0.5%. The upper eyelid is everted and the conjunctiva just superior to the upper tarsal edge is exposed. Using a 30-gauge needle, a single bolus of Hyaluronic Acid Gel is placed centrally in the subconjunctival levator-Muller plane. Small volumes (0.1 to 0.2 ml) of Hyaluronic Acid Gel are injected with the end point being adequate lowering with improved symmetry.
  Other Names: Restylane; Belotero
Drug: Saline injection — The conjunctiva is anesthetized with Proparacaine Hydrochloride Ophthalmic Solution, 0.5%. The upper eyelid is everted and the conjunctiva just superior to the upper tarsal edge is exposed. Using a 30-gauge needle, a single bolus of saline is placed centrally in the subconjunctival levator-Muller plane. Small volumes (0.1 to 0.2 ml) of saline are injected with the end point being adequate lowering with improved symmetry.
  Other Names: Normal saline

SUMMARY:
Thyroid eye disease (TED) is an autoimmune disease that affects the eye area. The disease presents with a variety of physical findings, including bulging of the eyes (proptosis), upper and lower eyelid retraction, and swelling/inflammation of the eye itself.

The disease passes through two phases: active and inactive. The active phase lasts between 18 and 24 months. During this phase, TED signs and symptoms generally worsen and then often improve. The inactive phase follows, during which the signs and symptoms of TED cease to improve and usually stabilize.

Lid retraction is a cardinal sign of TED. In addition to potentially causing cornea damage due to improper lid closure, lid retraction is also very troublesome for patients due to its cosmetic appearance. The precise pathophysiology of lid retraction is poorly understood, but a leading hypothesis is that it occurs due to scarring and fibrosis in the muscles that lift the eyelid.

Currently, the definitive treatment for lid retraction is surgery, which can be used to lengthen the lid itself or remove inflamed tissue from behind the eye, thus causing the eye to bulge less. In cases when patients first present to their physician with corneal ulceration or compression of the optic nerve, surgery may be performed immediately. However, in most instances, surgical procedures are delayed until the active stage of the disease has passed. Thus, most patients must endure the cosmetic and irritant symptoms of TED for up to two years.

Hyaluronic Acid Gels (HAG) have been FDA approved for the treatment of facial rhytids (wrinkles). They are injected under the skin and work by increasing volume. Recently, some smaller retrospective research studies have shown that HAG is also effective in correcting upper and lower eyelid retraction in TED. Hence, HAG may be for patients with active stage TED. It is also thought that if employed early in active phase disease, HAG may also help to decrease the severity of associated symptoms and reduce the need for surgery.

The purpose of the current investigation is to define the clinical utility of HAG correction of upper eyelid in active TED in terms of anatomic (lid position), quantitative (corneal dry eye signs) and qualitative effects (symptom severity and thyroid related quality of life).

ELIGIBILITY:
Inclusion Criteria:

1. Active stage TO as determined by symptom onset of under 9 months.
2. Upper eyelid retraction of 1mm or greater in one or both eyes.
3. Complaints of either significant ocular symptoms (despite appropriate use of ocular lubricants), or cosmetic deformity associated with the eyelid retraction.

Exclusion Criteria:

1. Age less than 21 years: due to lack of data on safety for HAG fillers in pediatric population
2. Age over 65 years of age: as HAG filler effect may be different in this population
3. Are pregnant or nursing: as there is little safety data on potential teratogenicity of HAG fillers
4. Have a demonstrated allergy to HAG fillers or lidocaine
5. Have a current infection, skin sore, pimple, rash, hive or cyst over the injection site: to avoid worsening the infection or transmitting it
6. Have a bleeding disorder or currently taking blood thinning medications such as Coumadin, heparin or acetylsalicylic acid on a daily basis.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-12; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Upper eyelid scleral show and marginal reflex distance 1 in mm | 6 weeks after injection
  Physicians will measure the amount of lid retraction (upper eyelid scleral show, marginal reflex distance 1) present in study participants 6 weeks following injection of hyaluronic acid gel vs. saline.

SECONDARY OUTCOMES:
Dry Eye | 6 weeks post injection.
  We will measure severity of dry eye signs using the Oxford staining scale and the Ocular surface disease index
Quality of life | 6 weeks
  The Graves Orbitopathy Quality of Life (GO-QOL) survey will be given to subjects at entry and at 6 weeks.
Complications | 6 weeks
  Complications including null effect, ecchymosis, retrobulbar hemorrhage, cranial nerve injury and extraocular muscle dysfunction will be monitored and reported

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rootman, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Jules Stein Eye Institute, Los Angeles, California
  - The Jules Stein Eye Institute at UCLA, Los Angeles, California